CLINICAL TRIAL: NCT04777526
Title: Clinical Effects of a Proprioceptive Thumb Exercise for Individuals With Carpometacarpal Joint Osteoarthritis: A Prospective Quasi-experimental Study
Brief Title: Effectiveness of Proprioceptive Exercises Program in Patients With Carpometacarpal Joint Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Raquel Cantero-Téllez, Clinical Professor, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-20
Record Dates: First submitted 2021-02-21; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Thumb Osteoarthritis
Keywords: Thumb pain; Thumb proprioception; Thumb Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Thumb orthosis at night. Daily exercises program during 4 weeks grouped in 3 sets of 10 repetitions in absence of pain. Exercises will consisted of active
  - resistive exercises for the first dorsal interosseous (FDI) muscle, manual distraction of the CMC joint and relaxation of the adductor thumb muscle.
  Interventions: Other: Joint protection program; Other: Thumb orthosis; Other: Manual distraction
- Experimental group (Experimental): The experimental group will also carried out a proprioceptive exercise program divided in three phases of 2 weeks per phase.
  Interventions: Other: Proprioception exercises; Other: Joint protection program; Other: Thumb orthosis; Other: Manual distraction

INTERVENTIONS:
Other: Proprioception exercises — Exercises for recognition of thumb position and thumb force sense.
  Arms: Experimental group
Other: Joint protection program — Reeducation in the activities daily life
Other: Thumb orthosis — Thumb night orthosis
Other: Manual distraction — Manual distraction of CMC joint

SUMMARY:
Objective: To establish the effectiveness of a proprioceptive training program as a complementary therapy for a traditional protocol in position control, pain intensity, upper limb function and occupation performance for patients with thumb CMC joint OA.

Methods: Standard conservative thumb CMC joint OA treatments were received for both the control (n=26) and experimental groups (n=26) for a period of 12 weeks. The experimental group received a proprioceptive training program during the same intervention period, which was conducted twice weekly (24 sessions). The severity of pain with activity was measured according to the visual analog scale (VAS). QuickDASH questionnaire was used to measure upper extremity function. Patient's occupational performance was measured with the Canadian Occupational Performance Measure (COPM) and proprioception was assessed using Joint position sense (JPS) testing.

ELIGIBILITY:
Inclusion Criteria:

Patients were included if they satisfied the following inclusion criteria; over 18 years of age with a diagnosis of grade I, II or III thumb CMC joint OA in their dominant hand according to the Eaton Classification Stage (14), a minimum pain rating of 4/10 on the Visual Analogue Scale (VAS) during activities of daily living (ADLs) at the time of the therapy initial evaluation,and the ability to read and understand the patient information sheets and exercises.

Exclusion Criteria:

Patients were excluded from participation if they had a neurological disorder affecting the upper limb, had received specific treatment for hand or thumb pain in the same limb in the last 6 months including an intra-articular joint injection to wrist, fingers, or thumb, had fractures or a significant hand injury or previous surgery to the wrist or hand, or had hand or finger tenosynovitis and/or Dupuytren disease. We also excluded patients with cognitive impairments who were not able to understand the informed consent and/or exercise program.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-07-18 (Actual)

PRIMARY OUTCOMES:
Joint position Sense (JPS) | 12 weeks
  Proprioception using active joint position sense (JPS) has been utilized in studies to establish a correlation between therapy intervention and proprioception. The target position of 30o CMC abduction will be selected. Joint angle will be measured using a standard clear plastic goniometer.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | baseline- 3- 12 weeks
  VAS has been shown to be a reliable and valid instrument for pain assessment which is used frequently for clinical and research purposes. It consists of a 10-cm line anchored at each end. The left-hand anchor reads 'no pain' and the right-hand anchor reads 'worst possible pain'; the patients marked a line to represent their pain level.
Canadian Occupational Performance Measure | baseline- 3- 12 weeks
  Patient's occupational performance will be measured with the Canadian Occupational Performance Measure (COPM). The COPM enables subjects to identify goals for hand therapy and engage in a subject-specific therapeutic process. It has been established that the COPM has good convergent validity and responsiveness for evaluating the relationship between patient self-perception and satisfaction for patients with CMC thumb OA .
Quick-dash | baseline- 3- 12 weeks
  The QuickDASH questionnaire will be used to measure upper extremity function. This tool consists of 11 items providing a total score ranging from 0 to 100 where 0 indicates no limitation and 100 suggests full disability. Eight items include questions about the ability of the patient to perform certain daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Cantero-Téllez, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No